CLINICAL TRIAL: NCT00471354
Title: Evaluation of Academic Performance in Asian Children Aged 8 to 11 Years With Attention-Deficit/Hyperactivity Disorder Treated With Atomoxetine Hydrochloride
Brief Title: A Study for Patients With Attention-Deficit/Hyperactivity Disorder Treated With Atomoxetine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, ELi Lilly
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11098; B4Z-CR-S018
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Results first posted 2009-12-31 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atomoxetine (Experimental): 0.5 mg/kg/day once a day (QD), by mouth (PO), starting dose titrated over 1 week to target dose 1.2 mg/kg/day QD, PO for 23 weeks.
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — atomoxetine 0.5 mg/kg/day once a day (QD), by mouth (PO) starting dose titrated over 1 week to target dose 1.2 mg/kg/day QD, PO for 23 weeks.
  Other Names: LY139603; Strattera

SUMMARY:
The purpose of the study is to investigate the relationship of changes in measures of academic performance and problem behaviors, to changes in core Attention-Deficit/Hyperactivity Disorder (ADHD) symptoms in Asian children treated with atomoxetine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients between 8 and 11 years of age at study entry
* Attention-Deficit/Hyperactivity Disorder (ADHD) meeting the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition, Text Revision (DSM-IV-TR) disease diagnostic criteria
* Patients who have never received medications psychotropic medications specifically to treat ADHD, or if they have received medication, that the trial of the psychotropic medication(s) was of less than 1 month duration, and occurred more than 6 months prior to study entry
* Normal intelligence in the judgment of the investigator
* Must be able to swallow capsules

Exclusion Criteria:

* Current or past history of bipolar I or II disorder, psychosis, autism, Asperger's syndrome, pervasive developmental disorder, or conduct disorder
* History of seizure disorder or currently taking anticonvulsants for seizure control
* Serious suicidal risk as determined by investigator
* Cardiovascular disease; current or past history of hypertension
* Previous treatment with atomoxetine

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 228 (Actual)
Dates: Start 2007-04; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- China (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Shanghai
- South Korea (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Pusan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Seoul
- Taiwan (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Neihu Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Niao Sung Hsiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Taipei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal ph, Taoyuan District

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Atomoxetine
Started | 228
Completed | 176
Not Completed | 52
Not completed — Protocol Entry Criteria Not Met | 1
Not completed — Adverse Event | 13
Not completed — Protocol Violation | 12
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 4
Not completed — Sponsor Decision | 1
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 5
Not completed — Patient/Caregiver Decision | 12

BASELINE CHARACTERISTICS:
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
Age Continuous [Mean (Standard Deviation); unit: years] | 9.6 (0.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 194
Region of Enrollment [Number; unit: participants]
  Taiwan | 76
  China | 82
  Korea, Republic of | 70
Diagnostic and Statistical Manual of Mental Disorders Fourth Edition Subtypes [Number; unit: participants]
  Hyperactive | 5
  Combined | 141
  Inattentive | 82
Race/Ethnicity [Number; unit: participants]
  East Asian | 228
Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS) Total Score [Mean (Standard Deviation); unit: units on a scale] — Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored - Total Score measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
  units on a scale | 35.3 (7.09)
Clinical Global Impression-Attention Deficit Hyperactivity Disorder-Severity Scale (CGI-ADHD-S) [Mean (Standard Deviation); unit: units on a scale] — Measures severity of the patient's overall severity of ADHD symptoms on a scale of 1-7 (1=normal, not at all ill; 7=among the most extremely ill patients).
  units on a scale | 5.0 (0.80)
Conners' Parent Rating Scale-Revised:Short Form - ADHD Index Subscale [Mean (Standard Deviation); unit: units on a scale] — A 27-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the parent to assess problem behaviors related to ADHD. ADHD Index score ranges from 0 to 36. Higher scores reflect more severe problem behaviors related to ADHD.
  units on a scale | 24.5 (5.90)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 136.4 (8.25)
School Grade Average (SGA) Language Score [Mean (Standard Deviation); unit: units on a scale] — Language school grade on a scale of 0-100, with higher scores indicating better grades/apptitude in language.
  units on a scale | 73.8 (18.35)
School Grade Average (SGA) Math Score [Mean (Standard Deviation); unit: units on a scale] — Math school grade on a scale of 0-100, with higher scores indicating better grades/apptitude in math.
  units on a scale | 72.7 (19.89)
School Grade Average (SGA) Total Score [Mean (Standard Deviation); unit: units on a scale] — School grades in the classes of Language, Math, and Science were obtained. A score between 0 and 100 was provided for each of the three classes, and the average taken to get a SGA Total Score between 0 and 100, with higher scores indicating better grades/apptitude.
  units on a scale | 73.9 (15.82)
School Grade Score (SGA) Science Score [Mean (Standard Deviation); unit: units on a scale] — Science school grade on a scale of 0-100, with higher scores indicating better grades/apptitude in science.
  units on a scale | 75.0 (17.04)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 33.3 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Change From Baseline and 24 Week Endpoint in Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent:Investigator-Administered and Scored (ADHDRS-IV-Parent:Inv) Total Score and School Grade Average (SGA)
Description: Correlation was calculated between change from baseline and endpoint in ADHD-RS Total Score and change in SGA total score. ADHD-RS measures 18 symptoms associated with diagnosis of ADHD. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. SGA: Grades (0 to 100) in classes of Language, Math, and Science were obtained and average taken to get SGA Total Score between 0 and 100; higher scores indicating better grades/apptitude. Any ordinal grades were imputed to numerical grades based on communication with relevant schools.
Time Frame: Baseline, 24 weeks
Population: All patients with baseline and at least one non-missing post-baseline score for each of the variables, regardless of them having or not having received any ordinal grades (for the SGA).
Measure: Number; unit: Spearman Correlation Coefficient
Arm/Group | Atomoxetine
Number analyzed (Participants) | 164
Spearman Correlation Coefficient | -0.083
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.293, Spearman Partial Rank Order Correlation

2. Secondary Outcome: Correlation Between Change From Baseline to 24 Week Endpoint in ADHDRS-IV-Parent:Inv Total Score and School Grade Averages in Separate Language, Math and Science Classes
Description: Correlation was calculated between change from baseline and endpoint in ADHD-RS Total Score and change in separate SGA language, math, and science scores. ADHD-RS measures 18 symptoms associated with diagnosis of ADHD. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54. SGA: separate language, math, and science school grades on a scale of 0-100, with higher scores indicating better grades/apptitude in the respective class. Any ordinal grades were imputed to numerical grades based on communication with relevant schools.
Time Frame: Baseline, 24 weeks
Population: as for outcome 1
Measure: Number; unit: Spearman Correlation Coefficient
Arm/Group | Atomoxetine
Number analyzed (Participants) | 164
Spearman Correlation Coefficient
  Correlation with Language Scores | -0.086
  Correlation with Math Scores | -0.126
  Correlation with Science Scores | -0.058
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.276, Spearman Partial Rank Order Correlation — P-value for Correlation with Language Scores
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.110, Spearman Partial Rank Order Correlation — P-value for Correlation with Math Scores
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p = 0.464, Spearman Partial Rank Order Correlation — P-value for Correlation with Science Scores

3. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Academic Performance by School Grade Average (SGA) Total, and Separate Language, Math, and Science Scores
Description: Separate school grades in the classes of Language, Math, and Science were obtained. A score between 0 and 100 was provided for each of the three classes, and the average taken to get a SGA Total Score between 0 and 100, with higher scores indicating better grades/apptitude in each class and overall. Any ordinal grades were imputed to numerical grades based on communication with relevant schools.
Time Frame: Baseline, 24 weeks
Population: All patients with baseline and at least one non-missing post-baseline score for each of the variables. Last observation carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 177
units on a scale
  Change from Baseline in Language Scores | 3.9 (13.35)
  Change from Baseline in Math Scores | 4.1 (16.58)
  Change from Baseline in Science Scores | 6.1 (14.98)
  Change from Baseline in Total Scores | 4.7 (10.68)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value for Change from Baseline in Language Scores
Statistical Analysis 2: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value for Change from Baseline in Math Scores
Statistical Analysis 3: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value for Change from Baseline in Science Scores
Statistical Analysis 4: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test — P-value for Change from Baseline in Total Scores

4. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Attention-Deficit/Hyperactivity Disorder Rating Scale-IV-Parent Version:Investigator-Administered and Scored - Total Score
Description: Measures the 18 symptoms contained in the DSM-IV diagnosis of Attention-Deficit/Hyperactivity Disorder. Individual item scores range from 0 (none/never or rarely) to 3 (severe/very often). Total scores range from 0 to 54.
Time Frame: Baseline, 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 205
units on a scale | -18.8 (9.27)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test

5. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Clinical Global Impressions - Attention-Deficit/Hyperactivity Disorder - Severity Scale (CGI-ADHD-S)
Description: Measures severity of the patient's overall severity of ADHD symptoms (1=normal, not at all ill; 7=among the most extremely ill patients).
Time Frame: Baseline, 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
units on a scale | -2.1 (1.25)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test

6. Secondary Outcome: CGI-ADHD-Improvement Scale (CGI-ADHD-I) at 24 Week Endpoint
Description: Measures total improvement (or worsening) of a patient's ADHD symptoms from the beginning of treatment (1=very much improved, 7=very much worsened).
Time Frame: 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 228
units on a scale | 2.3 (1.05)

7. Secondary Outcome: Change From Baseline to 24 Week Endpoint in Revised Conners' Parent Rating Scale: Short Form (CPRS-R:S) Attention-Deficit/Hyperactivity Disorder Index Score
Description: A 27-item rating scale (0 [not at all/never] to 3 [very much true/very often]) completed by the parent to assess problem behaviors related to ADHD. Subscale assessed: ADHD Index. ADHD Index is the sum of items 1, 5, 7, 10, 13, 15, 17, 19, 21, 23, 25, and 27. Subscale total scores range from 0 to 36. Higher scores reflect more severe problem behaviors related to ADHD.
Time Frame: Baseline, 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Atomoxetine
Number analyzed (Participants) | 204
units on a scale | -9.8 (7.94)
Statistical Analysis 1: Comparison: Atomoxetine; Test type: Superiority or Other; p < 0.001, Paired t-test

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 24 week overall study period.
Arm/Group | Atomoxetine
Serious Adverse Events (participants affected / at risk) | 1/228
Other Adverse Events (participants affected / at risk) | 175/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=228)
Hyperthyroidism (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atomoxetine (N=228)
Abdominal pain upper (Gastrointestinal disorders) | 15 (16)
Nausea (Gastrointestinal disorders) | 49 (57)
Vomiting (Gastrointestinal disorders) | 26 (32)
Fatigue (General disorders) | 25 (28)
Irritability (General disorders) | 20 (24)
Nasopharyngitis (Infections and infestations) | 15 (15)
Weight decreased (Investigations) | 16 (19)
Anorexia (Metabolism and nutrition disorders) | 55 (61)
Decreased appetite (Metabolism and nutrition disorders) | 74 (91)
Dizziness (Nervous system disorders) | 31 (36)
Headache (Nervous system disorders) | 29 (33)
Somnolence (Nervous system disorders) | 46 (54)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days